CLINICAL TRIAL: NCT04516655
Title: A Phase II， Single-arm Trail of Chidamide Combined With Rituximab and High-dose Methotrexate in Previously Untreated Patients With Primary Central Nervous System Lymphoma
Brief Title: A Phase II Trail of Chidamide ,Rituximab and Methotrexate in Lymphoma Patients
Acronym: C-R-HDMTX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fangfang Lv, MD, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-R-HDMTX
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Central Nervous System Lymphoma
MeSH Terms: interventions — Rituximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-R-MTX (Experimental): chidamide 20 mg biw PO day1-14 and rituximab 375 mg/m2 IV given on day 1 and methotrexate 3.5g/m2 IV given on day 2 of every 21-day cycle for 6 cycles
  Interventions: Drug: chidamide combined with rituximab and high-dose methotrexate

INTERVENTIONS:
Drug: chidamide combined with rituximab and high-dose methotrexate — chidamide 20 mg biw PO day1-14 and rituximab 375 mg/m2 IV given on day 1 and methotrexate 3.5g/m2 IV given on day 2 of every 21-day cycle for 6 cycles in untreated patients with primary central nervous system lymphoma

SUMMARY:
This study will evaluate the efficacy, safety and patient reported outcomes of chidamide 20 mg biw PO day1-14 and rituximab 375 mg/m2 IV given on day 1 and methotrexate 3.5g/m2 IV given on day 2 of every 21-day cycle for 6 cycles in untreated patients with primary central nervous system lymphoma.

The primary study endpoint will be complete response (CR) rate as assessed by the investigator. The hypothesis is previously untreated patients with primary central nervous system lymphoma could achieve a CR rate of 80% with C-R-HDMTX.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG Performance Status of 0, 1, or 2
2. Previously untreated patients with primary central nervous system lymphoma with pathologically confirm
3. At least one bi-dimensionally measurable lesion, defined as >1.0 cm in its longest dimension as measured by MRI
4. Signed written Informed Consent Form
5. hematologic function,defined as follows:

   * Hemoglobin ³ 9.0 g/dL without packed RBC transfusion during 14 days before first treatment
   * ANC ³ 1,000/µL
   * Platelet count ³ 80,000/µL
6. Adequate liver and kidney function function,defined as follows:

Serum AST and ALT≤ 2.5 *ULN ，Total bilirubin ≤ 1.5 * ULN Serum creatinine clearance ≥ 50 mL/min (using Cockcroft-Gault formula)

Exclusion Criteria:

1. Evidence of extracranial involvement (such as testis and breast) and secondary CNS involvement
2. Evidence of pleural fluid, ascites and pericardial effusion
3. History or presence of prolonged QTc interval in ECG, QTc interval>470ms in female and >450ms in male
4. History of other malignancy in 5 years
5. Positive test results for hepatitis C, HIV and RPR.
6. Positive test results for chronic hepatitis B infection (defined as positive hepatitis B surface antigen [HBsAg] serology) Patients with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative HBsAg) may be included if hepatitis B virus (HBV) DNA is less than 10E4 at the time of screening.
7. Pregnancy or lactation or intending to become pregnant during study
8. Prior organ transplantation
9. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at study enrollment or significant infections within 2 weeks before the start of Cycle 1.
10. Evidence of significant, uncontrolled, epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
CR rate | up to 18 weeks
  CR rate of the lesion of previously untreated patients with primary central nervous system lymphoma according to the international collaborative evaluation criteria for central nervous system lymphoma （2005）with Enhanced MRI every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Fangfang Lv, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gerstner ER, Batchelor TT. Primary central nervous system lymphoma. Arch Neurol. 2010 Mar;67(3):291-7. doi: 10.1001/archneurol.2010.3. PMID 20212226
- [Result] Batchelor TT. Primary central nervous system lymphoma: A curable disease. Hematol Oncol. 2019 Jun;37 Suppl 1:15-18. doi: 10.1002/hon.2598. PMID 31187523
- [Result] Batchelor T, Carson K, O'Neill A, Grossman SA, Alavi J, New P, Hochberg F, Priet R. Treatment of primary CNS lymphoma with methotrexate and deferred radiotherapy: a report of NABTT 96-07. J Clin Oncol. 2003 Mar 15;21(6):1044-9. doi: 10.1200/JCO.2003.03.036. PMID 12637469
- [Result] Chamberlain MC, Johnston SK. High-dose methotrexate and rituximab with deferred radiotherapy for newly diagnosed primary B-cell CNS lymphoma. Neuro Oncol. 2010 Jul;12(7):736-44. doi: 10.1093/neuonc/noq011. Epub 2010 Feb 8. PMID 20511181
- [Result] DeAngelis LM, Seiferheld W, Schold SC, Fisher B, Schultz CJ; Radiation Therapy Oncology Group Study 93-10. Combination chemotherapy and radiotherapy for primary central nervous system lymphoma: Radiation Therapy Oncology Group Study 93-10. J Clin Oncol. 2002 Dec 15;20(24):4643-8. doi: 10.1200/JCO.2002.11.013. PMID 12488408
- [Result] Gavrilovic IT, Hormigo A, Yahalom J, DeAngelis LM, Abrey LE. Long-term follow-up of high-dose methotrexate-based therapy with and without whole brain irradiation for newly diagnosed primary CNS lymphoma. J Clin Oncol. 2006 Oct 1;24(28):4570-4. doi: 10.1200/JCO.2006.06.6910. PMID 17008697
- [Result] Shah GD, Yahalom J, Correa DD, Lai RK, Raizer JJ, Schiff D, LaRocca R, Grant B, DeAngelis LM, Abrey LE. Combined immunochemotherapy with reduced whole-brain radiotherapy for newly diagnosed primary CNS lymphoma. J Clin Oncol. 2007 Oct 20;25(30):4730-5. doi: 10.1200/JCO.2007.12.5062. PMID 17947720
- [Result] Wieduwilt MJ, Valles F, Issa S, Behler CM, Hwang J, McDermott M, Treseler P, O'Brien J, Shuman MA, Cha S, Damon LE, Rubenstein JL. Immunochemotherapy with intensive consolidation for primary CNS lymphoma: a pilot study and prognostic assessment by diffusion-weighted MRI. Clin Cancer Res. 2012 Feb 15;18(4):1146-55. doi: 10.1158/1078-0432.CCR-11-0625. Epub 2012 Jan 6. PMID 22228634
- [Result] Gregory G, Arumugaswamy A, Leung T, Chan KL, Abikhair M, Tam C, Bajel A, Cher L, Grigg A, Ritchie D, Opat S. Rituximab is associated with improved survival for aggressive B cell CNS lymphoma. Neuro Oncol. 2013 Aug;15(8):1068-73. doi: 10.1093/neuonc/not032. Epub 2013 Mar 15. PMID 23502429
- [Result] Holdhoff M, Ambady P, Abdelaziz A, Sarai G, Bonekamp D, Blakeley J, Grossman SA, Ye X. High-dose methotrexate with or without rituximab in newly diagnosed primary CNS lymphoma. Neurology. 2014 Jul 15;83(3):235-9. doi: 10.1212/WNL.0000000000000593. Epub 2014 Jun 13. PMID 24928128
- [Result] Ly KI, Crew LL, Graham CA, Mrugala MM. Primary central nervous system lymphoma treated with high-dose methotrexate and rituximab: A single-institution experience. Oncol Lett. 2016 May;11(5):3471-3476. doi: 10.3892/ol.2016.4393. Epub 2016 Mar 30. PMID 27123138
- [Result] Omuro A, Correa DD, DeAngelis LM, Moskowitz CH, Matasar MJ, Kaley TJ, Gavrilovic IT, Nolan C, Pentsova E, Grommes CC, Panageas KS, Baser RE, Faivre G, Abrey LE, Sauter CS. R-MPV followed by high-dose chemotherapy with TBC and autologous stem-cell transplant for newly diagnosed primary CNS lymphoma. Blood. 2015 Feb 26;125(9):1403-10. doi: 10.1182/blood-2014-10-604561. Epub 2015 Jan 7. PMID 25568347
- [Result] Glass J, Won M, Schultz CJ, Brat D, Bartlett NL, Suh JH, Werner-Wasik M, Fisher BJ, Liepman MK, Augspurger M, Bokstein F, Bovi JA, Solhjem MC, Mehta MP. Phase I and II Study of Induction Chemotherapy With Methotrexate, Rituximab, and Temozolomide, Followed By Whole-Brain Radiotherapy and Postirradiation Temozolomide for Primary CNS Lymphoma: NRG Oncology RTOG 0227. J Clin Oncol. 2016 May 10;34(14):1620-5. doi: 10.1200/JCO.2015.64.8634. Epub 2016 Mar 28. PMID 27022122
- [Result] Song Y, Wen Y, Xue W, Zhang Y, Zhang M. Effect of rituximab on primary central nervous system lymphoma: a meta-analysis. Int J Hematol. 2017 Nov;106(5):612-621. doi: 10.1007/s12185-017-2316-z. Epub 2017 Sep 12. PMID 28900847
- [Result] Ferreri AJ, Reni M, Foppoli M, Martelli M, Pangalis GA, Frezzato M, Cabras MG, Fabbri A, Corazzelli G, Ilariucci F, Rossi G, Soffietti R, Stelitano C, Vallisa D, Zaja F, Zoppegno L, Aondio GM, Avvisati G, Balzarotti M, Brandes AA, Fajardo J, Gomez H, Guarini A, Pinotti G, Rigacci L, Uhlmann C, Picozzi P, Vezzulli P, Ponzoni M, Zucca E, Caligaris-Cappio F, Cavalli F; International Extranodal Lymphoma Study Group (IELSG). High-dose cytarabine plus high-dose methotrexate versus high-dose methotrexate alone in patients with primary CNS lymphoma: a randomised phase 2 trial. Lancet. 2009 Oct 31;374(9700):1512-20. doi: 10.1016/S0140-6736(09)61416-1. Epub 2009 Sep 18. PMID 19767089
- [Result] Abrey LE, Moskowitz CH, Mason WP, Crump M, Stewart D, Forsyth P, Paleologos N, Correa DD, Anderson ND, Caron D, Zelenetz A, Nimer SD, DeAngelis LM. Intensive methotrexate and cytarabine followed by high-dose chemotherapy with autologous stem-cell rescue in patients with newly diagnosed primary CNS lymphoma: an intent-to-treat analysis. J Clin Oncol. 2003 Nov 15;21(22):4151-6. doi: 10.1200/JCO.2003.05.024. PMID 14615443
- [Result] Colombat P, Lemevel A, Bertrand P, Delwail V, Rachieru P, Brion A, Berthou C, Bay JO, Delepine R, Desablens B, Camilleri-Broet S, Linassier C, Lamy T. High-dose chemotherapy with autologous stem cell transplantation as first-line therapy for primary CNS lymphoma in patients younger than 60 years: a multicenter phase II study of the GOELAMS group. Bone Marrow Transplant. 2006 Sep;38(6):417-20. doi: 10.1038/sj.bmt.1705452. PMID 16951691
- [Result] Illerhaus G, Muller F, Feuerhake F, Schafer AO, Ostertag C, Finke J. High-dose chemotherapy and autologous stem-cell transplantation without consolidating radiotherapy as first-line treatment for primary lymphoma of the central nervous system. Haematologica. 2008 Jan;93(1):147-8. doi: 10.3324/haematol.11771. PMID 18166803
- [Result] Cote GM, Hochberg EP, Muzikansky A, Hochberg FH, Drappatz J, McAfee SL, Batchelor TT, LaCasce AS, Fisher DC, Abramson JS, Armand P, Chen YB. Autologous stem cell transplantation with thiotepa, busulfan, and cyclophosphamide (TBC) conditioning in patients with CNS involvement by non-Hodgkin lymphoma. Biol Blood Marrow Transplant. 2012 Jan;18(1):76-83. doi: 10.1016/j.bbmt.2011.07.006. Epub 2011 Jul 13. PMID 21749848
- [Result] Ferreri AJM, Cwynarski K, Pulczynski E, Fox CP, Schorb E, La Rosee P, Binder M, Fabbri A, Torri V, Minacapelli E, Falautano M, Ilariucci F, Ambrosetti A, Roth A, Hemmaway C, Johnson P, Linton KM, Pukrop T, Sonderskov Gorlov J, Balzarotti M, Hess G, Keller U, Stilgenbauer S, Panse J, Tucci A, Orsucci L, Pisani F, Levis A, Krause SW, Schmoll HJ, Hertenstein B, Rummel M, Smith J, Pfreundschuh M, Cabras G, Angrilli F, Ponzoni M, Deckert M, Politi LS, Finke J, Reni M, Cavalli F, Zucca E, Illerhaus G; International Extranodal Lymphoma Study Group (IELSG). Whole-brain radiotherapy or autologous stem-cell transplantation as consolidation strategies after high-dose methotrexate-based chemoimmunotherapy in patients with primary CNS lymphoma: results of the second randomisation of the International Extranodal Lymphoma Study Group-32 phase 2 trial. Lancet Haematol. 2017 Nov;4(11):e510-e523. doi: 10.1016/S2352-3026(17)30174-6. Epub 2017 Oct 17. PMID 29054815
- [Result] Thiel E, Korfel A, Martus P, Kanz L, Griesinger F, Rauch M, Roth A, Hertenstein B, von Toll T, Hundsberger T, Mergenthaler HG, Leithauser M, Birnbaum T, Fischer L, Jahnke K, Herrlinger U, Plasswilm L, Nagele T, Pietsch T, Bamberg M, Weller M. High-dose methotrexate with or without whole brain radiotherapy for primary CNS lymphoma (G-PCNSL-SG-1): a phase 3, randomised, non-inferiority trial. Lancet Oncol. 2010 Nov;11(11):1036-47. doi: 10.1016/S1470-2045(10)70229-1. Epub 2010 Oct 20. PMID 20970380
- [Result] Mohile NA, Deangelis LM, Abrey LE. The utility of body FDG PET in staging primary central nervous system lymphoma. Neuro Oncol. 2008 Apr;10(2):223-8. doi: 10.1215/15228517-2007-061. Epub 2008 Feb 20. PMID 18287338
- [Result] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Result] Yang H, Li C, Chen Z, Mou H, Gu L. Determination of chidamide in rat plasma and cerebrospinal fluid. Regul Toxicol Pharmacol. 2018 Oct;98:24-30. doi: 10.1016/j.yrtph.2018.07.001. Epub 2018 Jul 6. PMID 30008379
- [Result] Abrey LE, Batchelor TT, Ferreri AJ, Gospodarowicz M, Pulczynski EJ, Zucca E, Smith JR, Korfel A, Soussain C, DeAngelis LM, Neuwelt EA, O'Neill BP, Thiel E, Shenkier T, Graus F, van den Bent M, Seymour JF, Poortmans P, Armitage JO, Cavalli F; International Primary CNS Lymphoma Collaborative Group. Report of an international workshop to standardize baseline evaluation and response criteria for primary CNS lymphoma. J Clin Oncol. 2005 Aug 1;23(22):5034-43. doi: 10.1200/JCO.2005.13.524. Epub 2005 Jun 13. PMID 15955902